CLINICAL TRIAL: NCT03690258
Title: The Effects of Variable Load Exercise on Muscle Function and Blood Pressure Regulation: a Randomized Controlled Trail
Brief Title: Effects of Variable Load Exercise on Aging Atrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Split (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Damir Zubac, PhD, University Hospital of Split
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: ARRS: Z7-9420
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Sarcopenia; Hypertension; Muscle Atrophy
Keywords: muscle function; muscle fibers; systolic blood pressure
MeSH Terms: conditions — Sarcopenia; Hypertension; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Variable load exercise, non-pharmacological intervention
Who Masked: Investigator
Masking Description: Researches collecting data will be blinded of participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Variable load exercise (Experimental): Variable load intervention (The nHANCE-squat ultimate - iso-inertial load, with power output in watts performed 3 x per week) will being performed to determine whether this training approach is an effective countermeasure to attenuate for rapid declines in muscle power, function, contractile capacity that typically originate from aging and muscle disuse. Since age-related decline is accelerated already after short bouts of physical inactivity, with small recovery potential, any attempt to counteract age-related and disuse-related decline have high clinical significance. Based on the findings, we could develop safety guidelines and protocols aimed at reducing health risks in seniors.
  Data available at: http://nhance.se/
  Interventions: Device: Variable load exercise
- Variable load intervention (Experimental): This study is being conducted to determine whether this variable load (The nHANC dead lift - eccentric overload performed 3 x per week for 4-6 weeks) intervention is an effective countermeasure to modulate blood pressure in seniors. Since age-related incline in resting blood pressure (hypertension) is accelerated already after short bouts of physical inactivity, any attempt to counteract age-related and disuse-related decline have high clinical significance. In addition, we aim to examine endothelial function via non-invasive flow mediated dilatation (FMD) technique.
  Based on the findings, we could develop safety guidelines and protocols aimed at reducing health risks in this specific population. Importantly, in case present hypotheses are confirmed, this may offer important information to the healthcare system, especially for reducing economic burden.
  Interventions: Device: Variable load exercise

INTERVENTIONS:
Device: Variable load exercise — This study is being conducted to determine whether variable load training approach (nHANCE™ squat - more data available at http://nhance.se/) is an effective countermeasure to attenuate for rapid declines in muscle power, function, that typically originate from aging and muscle disuse. Since age-related decline is accelerated already after short bouts of physical inactivity, with small recovery potential, any attempt to counteract age-related and disuse-related decline have high clinical significance. Based on the findings, safety guidelines and protocols could be developed aimed at reducing health risks in seniors. Importantly, in case present hypotheses are confirmed, this may offer important information to the healthcare system.

SUMMARY:
The primary aim of this research proposal is to examine whether this novel training program approach is capable to tackle excessive loss in muscle mass, function and contractile capacity with aging. Previous investigations have universally shown a dramatic loss in type II muscle fibers, while certain countermeasures in their follow-up studies were generally ineffective and limited to attenuate this phenomenon. Probably, they failed to meet recruitment threshold of larger motor units and subsequently innervate type II muscle fibers. Furthermore, previous investigations also failed to provide any data on specific blood markers that may provide additional insight into muscle fiber loss with aging. Muscle fibers type II play a crucial role in the human ability to produce as much as force as possible over a limited time-frame (e.g. 100-200 ms) to counteract unexpected perturbations during stair climbing for example and thus avoiding falls. Therefore, this data collection would be noteworthy in particular, especially for this population due to health-related outcomes and healthy aging process.

Since age-related decline is accelerated already after short bouts of physical inactivity, with small recovery potential, any attempt to counteract age-related and disuse-related decline have high clinical significance. Based on the findings, data collected may aid in development of safety guidelines and protocols aimed at reducing health risks in this specific population. Importantly, in case the aforementioned hypotheses are confirmed, present findings may offer important information to the healthcare system, especially for reducing economic burden.

DETAILED DESCRIPTION:
This study is being conducted to determine whether a novel training approach (variable load exercise) is an effective countermeasure to attenuate for rapid declines in muscle power, function, contractile capacity and fiber type distribution that typically originate from aging and muscle disuse.

The present study is planned over a 24-month investigation period, including ethics application write-up, equipment calibration, participant recruitment, general health examination, familiarization trails, pilot study, data collection in the main portion of the study, data analysis and paper write-up for peer-review journal.Collaboration with Institute for Kinesiology Research of Koper (a municipality in Slovenia), University of Split, University of Udine and Padua is planned. In addition, recruitment of students of Applied Kinesiology at University of Primorska, to collaborate on data collection so they could use data acquired to write their final papers or master thesis is also planned.

After obtaining ethical approval, seniors will be recruited from the Primorska region in Slovenia, via presentations in Daily Activity Centers, social medial and local newspaper. Exclusion and inclusion criteria will be applied as outlined in the next paragraph and those applicants remaining will be randomized into different groups. Data collection will be carried out on eight separate occasions, including familiarization, pilot testing, main portion of the study and follow up data collection, in a randomized counter balance crossover fashion. Following familiarization and pilot study all participants will be randomly assigned to either (I) RT or (II) variable load exercise (VLE) before a crossover of experimental protocols is executed, after a minimum washout period (2x times the duration of experimental protocol) and a follow-up measurement will take place two weeks after experimental protocols are completed. Each participant will be allocated into RT or VLE with pre/post measurements preceding each condition, for eight consecutive weeks following a structured linear periodization model, previously used in healthy older adults (Colon et al., 2017). In total of 2 weeks of familiarization period (to ensure reliability of assessment and avoid learning effects), 4 weeks of pilot study (comparing old and young participants) 16 weeks of different training protocols (RT and VLE, plus 4 weeks of washout period) accompanied with follow-up measurements two weeks after completing training protocols, since training effects are in general dose-dependent and their effects are reversible. Lastly, testing procedures will be conducted at the same facility, by the same researchers using the same equipment at the similar time of the day across the investigation.

The selection of participants will consist of both male and female adults established on a purely voluntary basis. We will follow a strict inclusion and exclusion criteria (in brief):

1. Inclusion criteria: (Signed informed consent and doctor's permission; Age >50 years)
2. Exclusion criteria: (Any cardiovascular disease or ECG examination abnormalities (at rest and under load); hypertension (resting BP > 140/90 mm Hg); previous history of musculoskeletal and neurological disorder/injury; previous history of neurological disorders; supplement or drug consumption that may interfere with training outcomes; alcohol consumption and smoking; BMI >30 kg/m2).

The risks and benefits will be outlined to each participant before inclusion into the study. Risks include potential transient discomfort from the venipuncture blood sampling and muscle soreness originating from experimental training protocols. The participants will get valuable information on how their muscles adapt following systematic training protocols.

Experimental Protocol (Total experimental time: ~120 min for all trails, pre/post data collection):

1. Arrival to laboratory, anthropometric characteristics assessment; resting BP measurement
2. Rest, supine 30 min; complete blood sampling to measure inflammation response;
3. Perform non-invasive muscle composition assessment with Tensiomyography (TMG) of lower limbs;
4. Perform high density surface electromyography (HD EMG) of vastus lateralis and medialis muscles;
5. Perform muscle architecture assessment by ultrasound imaging;
6. Perform muscle voluntary contractions using dynamometry .
7. Energy cost of locomotion assessment

In order to increase the accuracy of the results of the study, all individuals will participate in a two session familiarization period before the study began. The subjects were asked to withdraw from intense physical activity two days prior to baseline assessment. All assessments will be performed in a closed and ventilated facility, with a temperature range of 18-22 C during the morning, and by the same researchers.

Intervention: To determine the optimal load during a single training session of multiple joint squat exercise by using the flywheel (FW) device (http://nhance.se/products/nhance-squat-ultimate/). A large number of papers were published in this area demonstrating that this sort of eccentric muscle overload is beneficial in terms of muscle power gains, balance improvements, contractile capacity, early architecture changes etc., in aging population. The key advantage of this sort of exercise (compared to classical RT) is that this device is equipped with three different wheels, providing different inertia (load), corresponding to 0.025, 0.05, 0.1 kg m2. Even more, this device offers an actual power output feedback (in Watts) in real-time. Thus, this allows us to benchmark a certain threshold where actual changes in both neuromuscular and cardiovascular system(s) occur (in case of continuous BP monitoring, of course) occur.

The originality of the expected results - A large number of recently published papers were looking at different modalities of RT with constant loads, different periodization models and their effects on muscle recovery in this specific population. However, their findings clearly showed that regardless of RT training or different training periodization strategies type II muscle fibers kept declining with muscle disuse and aging. Thus, one could speculate that sudden mechanical overload approach (or variable iso-inertial load) will be a viable tool to tackle muscle power and function loss via additional type II muscle fibers recruitment patterns. In addition, the present study aims to determine whether some specific blood markers (like agrin) could detect neuromuscular junction alterations following these experimental protocols.

ELIGIBILITY:
1. Inclusion criteria:

   Both genders will be included;
   * signed informed consent and doctor's permission;
   * Age >50 years;
   * BMI <30 kg/m2,
   * At least 30 minutes of daily moderate-to-vigorous physical activity during (including five days of monitoring prior to any data collection).
2. Exclusion criteria:

   * Severe cardiovascular diseases;
   * hypertension prevalence (>140/90 mm Hg).
   * history of severe musculoskeletal and neurological disorders/injuries;
   * history of severe neurological disorders;
   * supplement or drug consumption that may interfere with training outcomes;
   * alcohol consumption and smoking;
   * use of walking aids;

The risks and benefits will be outlined to each participant before inclusion into the study.

Data collection risks include potential transient discomfort from the venipuncture blood sampling and muscle soreness originating from experimental training protocols. The participants will get valuable information on how their muscles adapt following systematic training protocols.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Continuous blood pressure monitoring via photopletismograpy (via Finometer) and non-invasive hemodynamics assessment | 12-24 months
  Non-pharmacological intervention (exercise intervention); To address motor unit recruitment pattern with pre-post intervention data collection scheme.
Non invasive surface electromyography (HD EMG, in mV) during MVC (maximal voluntary contraction, Nm), Peak oxygen uptake assessment (VO2; ml kg min-1) | 12-24 months
  Pulmonary ventilation and oxygen uptake at rest and during cycling. All data will be collected via a portable system (K5 RQ, Cosmed, Rome, Italy)

SECONDARY OUTCOMES:
Endothelial function (via non invasive flow mediated dilatation technique | 12-24 months
  During exercise testing we plan to use s it is a portable ultrasound imaging

CONTACTS AND LOCATIONS:
Overall Officials: Rado Pisot, PhD, Study Director — Science and Research Center Koper, Institute for Kinesiology Research
Locations (2):
- Slovenia (2):
  - University of Primorska, Koper
  - ZRS Koper, Koper

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zubac D, Obad A, Ivancev V, Valic Z. Acute flywheel exercise does not impair the brachial artery vasodilation in healthy men of varying aerobic fitness. Blood Press Monit. 2021 Jun 1;26(3):215-223. doi: 10.1097/MBP.0000000000000523. PMID 33590994
- See also: Related Info — http://www.zrs-kp.si/